CLINICAL TRIAL: NCT02019303
Title: Ultrasound Guided Core Needle Biopsy Versus Fine Needle Aspiration of Morphologically Abnormal Axillary Lymph Node in Patients With New Diagnosis or Suspected Diagnosis of Invasive Breast Carcinoma
Brief Title: Accuracy of FNA Versus CNB of Abnormal Axillary Lymph Nodes in Setting of Invasive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Nicole Winkler, M.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 00068472
Record Dates: First submitted 2013-12-03; First posted 2013-12-24 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abnormal lymph nodes (Other): There is only one arm to this study and includes all eligible and consented patients with abnormal axillary lymph node on ultrasound.
  Interventions: Procedure: FNA and Core biopsy

INTERVENTIONS:
Procedure: FNA and Core biopsy — Both procedures will be performed on the same lymph node

SUMMARY:
To compare accuracy of ultrasound guided fine needle aspiration (FNA) to core needle biopsy (CNB) of ultrasound detected abnormal axillary lymph nodes in patients with newly diagnosed invasive breast cancer or suspected invasive breast cancer.

Hypothesis: FNA and CNB have equivalent diagnostic accuracies

In order to prove our hypothesis, we will perform FNA and CNB on the same lymph node in each consented patient. The two samples will be evaluated separately by different pathologists blinded to the material in the other sample.

The results of the biopsies will be compared to the gold standard (lymph node excision).

ELIGIBILITY:
Inclusion Criteria:

* Recent or suspected diagnosis of invasive breast cancer with abnormal ipsilateral axillary lymph node
* Able to provide informed consent

Exclusion Criteria:

* Lymph node not amenable to core biopsy
* Patient is unlikely to undergo lymph node excision (i.e. elderly patient with co-morbidities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of FNA and CNB | 2 years
  Accuracy will be determined by comparing the results of the FNA and CNB performed on the same lymph node to the gold standard using a paired test of equivalence. The gold standard is the final pathologic diagnosis of excised lymph node containing biopsy marker (either sentinel lymph node biopsy or axillary dissection). Surgical excision of pre-operatively sampled lymph node marks the end of study participation for each patient.

SECONDARY OUTCOMES:
Pain associated with FNA and CNB | 2 years
  Pain associated with each biopsy method will be assessed with a visual analog scale (0- 10) after a baseline pain measurement. The results will be compared to baseline pain level and analyzed using a paired t test.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Hospital, Salt Lake City, Utah, United States